CLINICAL TRIAL: NCT02189486
Title: Biomarkers and Clinical Parameters Associated With Gleason Score Upgrading
Brief Title: Prostate Cancer Upgrading Reference Set
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Emory University (Other); Stanford University (Other); University of California, Irvine (Other); University of Michigan (Other); The Cleveland Clinic (Other); University of Washington (Other); Fred Hutchinson Cancer Center (Other); University of Miami (Other); Johns Hopkins University (Other); M.D. Anderson Cancer Center (Other); Weill Medical College of Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other); Eastern Virginia Medical School (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSC20140367H; 5P30CA054174 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-14 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Prostate biopsy; Upgrading; Upgrading Reference set
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, voided urine and prostate tissue slides and blocks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prostate Cancer Cohort: Men with prostate cancer who have elected radical prostatectomy for their treatment of their prostate cancer within two years after prostate biopsy.

SUMMARY:
Research repository designed to establish prostate cancer upgrading reference set and development of a risk prediction tool. Repository will include clinical information and biologics on a cohort of 240 men, to predict presence of high grade cancer at time of prostatectomy (removal of prostate) among patients with a low grade cancer diagnosis at time of biopsy.

DETAILED DESCRIPTION:
The primary endpoint of this study is the presence of tumor upgrading at the time of radical prostatectomy. Upgrading is defined as: Gleason 3+4 or higher grade A secondary study endpoint is presence of prostate cancer beyond the prostate (pathologic T3 disease) at radical prostatectomy. (This finding may be considered as a rationale for treatment.) Evidence of pathologic stage T3 or higher disease will be assessed by the presence of: (1) seminal vesicle invasion or (2) positive surgical margins or (3) established extracapsular extension or (4) lymph node involvement by tumor. It should be noted that pathologic stage T3 disease, while generally portending a greater risk of disease recurrence, may not be an intrinsic feature of disease prognosis but can be an artifact of surgical technique. Nonetheless, a secondary risk assessment tool will include both a Gleason 7-10 endpoint plus any patients with pT3+ disease to a composite endpoint that could indicate disease best managed with treatment in lieu of active surveillance.Prostate cancer, confirmed on prostate biopsy, within two years of scheduled radical prostatectomy.

2. Prostate cancer must be graded as Gleason 3+3 on the biopsy immediately prior to radical prostatectomy. (Secondary eligibility will be established on central review of pathology slides, and blocks if available, at Cornell Central Pathology Laboratory to confirm eligibility.) 3. Prostate cancer may have been detected on prior biopsy as well but must not be greater than Gleason 3+3. (Also requires Central Pathology Laboratory review.) 4. Slides must be available for Central Pathology Laboratory review on any biopsy showing prostate cancer. FFPE (formalin fixed paraffin embedded) blocks may also be requested if available.

5. Patient must have selected radical prostatectomy as treatment for prostate cancer.

6. Signed informed consent. 7. Blocks and/or slides from prostate biopsy and from radical prostatectomy must be available for analysis by Central Pathology laboratory.

8. Willingness to provide long-term follow-up information regarding additional treatments and cancer status.

9. Willingness to provide blood and urine specimens prior to radical prostatectomy for placement in the Early Detection Research Network (EDRN) Upgrading Reference Set repository.

10. Willingness to provide demographic and clinical information related to prostate cancer and prostate cancer risk (e.g., race/ethnicity, family history of prostate cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer, confirmed on prostate biopsy, within two years of scheduled radical prostatectomy.
2. Prostate cancer must be graded as Gleason 3+3 on the biopsy immediately prior to radical prostatectomy. (Secondary eligibility will be established on central review of pathology slides, and blocks if available, at Cornell Central Pathology Laboratory to confirm eligibility.)
3. Prostate cancer may have been detected on prior biopsy as well but must not be greater than Gleason 3+3. (Also requires Central Pathology Laboratory review.)
4. Slides must be available for Central Pathology Laboratory review on any biopsy showing prostate cancer. FFPE Blocks may also be requested if available.
5. Patient must have selected radical prostatectomy as treatment for prostate cancer.
6. Signed informed consent.
7. Blocks and/or slides from prostate biopsy and from radical prostatectomy must be available for analysis by Central Pathology laboratory.
8. Willingness to provide long-term follow-up information regarding additional treatments and cancer status.
9. Willingness to provide blood and urine specimens prior to radical prostatectomy for placement in the EDRN Upgrading Reference Set repository.
10. Willingness to provide demographic and clinical information related to prostate cancer and prostate cancer risk (e.g., race/ethnicity, family history of prostate cancer).

Exclusion Criteria:

1. Gleason score greater than 3+3 on any prior prostate biopsy.
2. Any treatment other than radical prostatectomy planned for prostate cancer.
3. Prior treatment of the prostate with androgen deprivation, radiation, or other cytotoxic chemotherapy.

Ages: 35 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit a cohort of 600 men with prostate cancer who have elected radical prostatectomy for treatment of their prostate cancer within two years after prostate biopsy. This biopsy must show no greater grade than Gleason 3+3 disease as determined on central pathology review. The patient may have had previous biopsies that showed cancer but may never have had a tumor grade greater than Gleason 3+3.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2014-08; Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Prostate cancer tumor upgrading at time of radical prostatectomy (Gleason 3+4 or higher grade) | 4 years
  The primary endpoint of this study is the presence of tumor upgrading at the time of radical prostatectomy. Upgrading is defined as: Gleason 3+4 or higher grade

SECONDARY OUTCOMES:
Presence of prostate cancer beyond the prostate at radical prostatectomy (pathologic T3 disease) | 10 years
  A secondary study endpoint is presence of prostate cancer beyond the prostate (pathologic T3 disease) at radical prostatectomy. (This finding may be considered as a rationale for treatment.) Evidence of pathologic stage T3 or higher disease will be assessed by the presence of: (1) seminal vesicle invasion or (2) positive surgical margins or (3) established extracapsular extension or (4) lymph node involvement by tumor. It should be noted that pathologic stage T3 disease, while generally portending a greater risk of disease recurrence, may not be an intrinsic feature of disease prognosis but can be an artifact of surgical technique. Nonetheless, a secondary risk assessment tool will include both a Gleason 7-10 endpoint plus any patients with pT3+ disease to a composite endpoint that could indicate disease best managed with treatment in lieu of active surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Thompson Jr, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States